CLINICAL TRIAL: NCT04773106
Title: Follow-up of the First in Man, Prospective, Open-label, Single Arm, Multicenter Clinical Investigation to Assess the Long-term Safety and Performance of the ARGOS-SC Suprachoroidal Pressure Sensor System in Patients With Glaucoma Underwent Non-penetrating Glaucoma Surgery (Follow-up Month 12 - Month 36)
Brief Title: Long-term Safety and Performance of the ARGOS-SC Suprachoroidal Pressure Sensor System in Patients With Glaucoma Underwent Non-penetrating Glaucoma Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implandata Ophthalmic Products GmbH (Industry)
Collaborators: CRO Dr. med Kottmann GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARGOS-SC01_Follow-up; CIV-19-11-030784 (Registry Identifier: Eudamed)
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma; Open Angle Glaucoma
Keywords: Non-penetrating glaucoma surgery; Open angle glaucoma; Intraocular pressure measurements; Suprachoroidal pressure sensor; ARGOS-SC
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARGOS-SC Sensor (Other): The ARGOS-SC sensor was already implanted in the earlier ARGOS-SC01 study.
  Interventions: Device: ARGOS-SC suprachoroidal pressure sensor

INTERVENTIONS:
Device: ARGOS-SC suprachoroidal pressure sensor — The ARGOS-SC pressure sensor was additionally implanted during routine local intraocular pressure lowering procedures in patients with glaucoma undergoing non-penetrating glaucoma surgery in the earlier ARGOS-SC01 study.
  Other Names: EYEMATE-SC

SUMMARY:
The purpose of this study is to evaluate the long-term safety and performance of the ARGOS-SC system.

DETAILED DESCRIPTION:
This study is designed as a prospective, open-label, multicenter, single-arm clinical investigation. This study is a follow-up study to the ARGOS-SC01 study (NCT03756662). Patients who have graduated the ARGOS-SC01 study after 12 month follow-up will be asked to enroll in this study for an additional 24 month follow-up (month 12-36 post implantation). This study will be solely observational, as only patients who had implanted the device within the earlier study will be invited to join this ARGOS-SC01_FU study.

The sensor was always implanted in one eye only which will be the study eye.

ELIGIBILITY:
Inclusion Criteria:

- Subjects of the ARGOS-SC01 study with an implanted ARGOS-SC suprachoroidal pressure sensor.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szurman, Prof., Principal Investigator — Knappschaftsklinikum Saar GmbH
Locations (5):
- Germany (4):
  - Universitäts-Augenklinik Bochum, Bochum
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Augenklinik und Poliklinik, Mainz
  - Augenklinik der LMU München, München
  - Knappschaftsklinikum Saar GmbH, Augenklinik Sulzbach, Sulzbach
- Swiss Glaucoma Research Foundation, Centre du Glaucome, Clinique Montchoisi, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Micheletti E, Mansouri K, Dick HB, Hoffmann EM, Mackert MJ, Weinreb RN, Szurman P; EYEMATE-SC Study Group. Long-term Safety and Performance of a Suprachoroidal Pressure Sensor System: Results of the EYEMATE-SC Trial Follow-up Study. Ophthalmology. 2025 Jul;132(7):775-784. doi: 10.1016/j.ophtha.2025.01.021. Epub 2025 Jan 31. PMID 39892748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from December 2019 to February 2021 in medical clinics.
Pre-assignment Details: Of the ARGOS-SC01 subjects, 22 patients consented to the ARGOS-SC01 follow-up study.
Groups:
- ARGOS-SC Sensor: ARGOS-SC pressure sensor previously implanted in the ARGOS-SC01 study during routine local intraocular pressure lowering procedures in patients with glaucoma undergoing non-penetrating glaucoma surgery.
  ARGOS-SC system: An active implantable intraocular pressure sensor implanted in the suprachoriodal space of the human eye, in combination with non-penetrating glaucoma surgery.
Period: Overall Study
Arm/Group | ARGOS-SC Sensor
Started | 22
Completed (Of the 22 patients enrolled, three patients voluntarily withdrew from the study during the follow-up and one patient deceased for unrelated reasons.) | 18
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All ARGOS-SC01 patients who have consented to the ARGOS-SC01 follow-up study.
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 4
  Germany | 18
Type of Glaucoma [Count of Participants; unit: Participants]
  Primary open-angle glaucoma (POAG) | 15
  Ocular hypertension (OHT)/Glaucoma suspect | 2
  Pseudoexfoliative (PEX) glauoma | 2
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Performance: Level of Agreement Between GAT and the ARGOS-SC System
Description: Level of Agreement between intraocular pressure (IOP) measurements made using GAT & the ARGOS-SC system (IOP in mmHg) following the Bland-Altman method.
Time Frame: Day 360 to Day 1080 (V09 to V13)
Population: All available GAT and ARGOS-SC measurements.
Measure: Mean (95% Confidence Interval); unit: mmHg
Units Other Than Participants: measurements
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 22
Number analyzed (measurements) | 522
mmHg | -0.3 [-6.2 to 5.7]

2. Secondary Outcome: Safety: Number of Patients Experiencing a Device-related SAE (SADE)
Description: Number of patients experiencing a device-related SAE (SADE)
Time Frame: Day 360 to Day 1080 (V09 to V13)
Measure: Count of Participants; unit: Participants
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 22
Participants | 0

3. Secondary Outcome: Safety: Incidence, Nature, Severity and Seriousness of Observed Adverse Events (AEs) and Adverse Device Events (ADEs)
Description: Safety evaluation based on the incidence, nature, severity and seriousness of observed adverse events and adverse device events.
Time Frame: Day 360 to Day 1080 (V09 to V13)
Population: A total of 50 AEs in 16 patients were reported in the ARGOS-SC follow-up study. In overall 15 adverse events were documented in 14 patients affecting the study eye. 12 out of 50 AEs in 7 patients fulfilled at least one criterion for "serious adverse event" (SAE) and were reported as such. All of these SAEs were unrelated to the medical device.
Measure: Number; unit: A(D)Es
Units Other Than Participants: Total number of AEs
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 16
Number analyzed (Total number of AEs) | 50
A(D)Es
  Overall number of AEs/ADEs | 50
  Overall number of AEs/ADEs affecting the study eye, of which: number analyzed (Participants) | 14
  Overall number of AEs/ADEs affecting the study eye, of which: number analyzed (Total number of AEs) | 15
  Overall number of AEs/ADEs affecting the study eye, of which | 15
  AEs related to medical procedure and/or: number analyzed (Participants) | 1
  AEs related to medical procedure and/or: number analyzed (Total number of AEs) | 15
  AEs related to medical procedure and/or | 1
  AEs related to medical device and/or: number analyzed (Participants) | 1
  AEs related to medical device and/or: number analyzed (Total number of AEs) | 15
  AEs related to medical device and/or | 1
  AEs related to other: number analyzed (Participants) | 6
  AEs related to other: number analyzed (Total number of AEs) | 15
  AEs related to other | 7

4. Secondary Outcome: Performance: Percentage of Measurements Within +/- 5 mmHg
Description: Concordance of the ARGOS-SC<>GAT measurement. Method applied: The probability distribution of the difference in the measurements made using GAT & the ARGOS-SC system per visit ("paired measurement") grouped within 1 mmHg was compared to the outcome measure of achieving 65% agreement of the total number of comparisons between +/-5 mmHg.
Time Frame: Day 360 to Day 1080 (V09 to V13)
Population: All available GAT<>ARGOS-SC comparisons.
Measure: Number; unit: percentage of comparisons
Units Other Than Participants: comparisons
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 22
Number analyzed (comparisons) | 86
percentage of comparisons | 94

5. Secondary Outcome: Performance: Device Malfunctions
Description: The number of observed device malfunctions / deficiencies (DDs) related to the ARGOS-SC system, consisting of the ARGOS-SC implant and an external handheld reader device for the activation, power supply, and readout of the implanted sensor.
Time Frame: Day 360 to Day 1080 (V09 to V13)
Population: Of the 22 patients, device deficiencies (all related to the Reader device (external handheld device)) have been documented for 10 patients, hence the 10 participants analyzed.
Measure: Number; unit: DDs
Units Other Than Participants: DDs
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 10
Number analyzed (DDs) | 13
DDs | 13

6. Secondary Outcome: Usability: User Acceptance at the Investigational Site
Description: User acceptance of the ARGOS-SC system at the investigational site by means of evaluation of Investigator's questionnaires on a scale of 1 to 7 how strongly they agree to given statements (1 = totally disagree, 7 = totally agree). Overall Number of Participants Analyzed represents the 8 physician investigators who completed the User Acceptance Questionnaire. The score 7 represents a greater user acceptance.
Time Frame: Day 1080 (V13)
Population: The user acceptance questionnaire for physicians was collected from 8 investigators.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 8
score on a scale | 4.7 (3.9)

7. Secondary Outcome: Usability: User Acceptance at Home
Description: User acceptance of the ARGOS-SC system at home by means of evaluation of patient questionnaires on a scale of 1 to 7 how strongly they agree to given statements (1 = totally disagree, 7 = totally agree). The score 7 represents a greater user acceptance.
Time Frame: Day 1080 (V13)
Population: Each patient was asked to provide feedback on the user acceptance of the ARGOS-SC system at home. A total of 15 patients provided feedback via a structured questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 15
score on a scale | 5.6 (3.6)

ADVERSE EVENTS:
Time Frame: Day 360 to Day 1080 (V09 to V13). In Germany the term SAE is defined according to §2 Section 5 MPSV.
Description: SAE defined as AE that
  1. Led to death
  2. Led to a serious deterioration in health of a subject that:
     a Resulted in life-threatening illness or injury b Resulted in permanent impairment of body-structure or function c Required in-patient hospitalization or prolongation of existing hospitalization d Required medical or surgical intervention to prevent permanent impairment to body-structure or a -function
  3. Led to foetal distress, foetal death or a congenital abnormality or birth defect
Arm/Group | ARGOS-SC Sensor
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 7/22
Other Adverse Events (participants affected / at risk) | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGOS-SC Sensor (N=22)
Bone fracture, upper arm (Injury, poisoning and procedural complications) | 1 (1)
Cardiac stent implantation (Surgical and medical procedures) | 1 (1)
Death, non-related (General disorders) | 1 (1)
Gastroenterological complaints (Gastrointestinal disorders) | 1 (1)
Hospitalization b/o nose surgery (removal of polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intestinal inflammation (Infections and infestations) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1)
Pain and fluid accumulation in the abdominal cavity (Gastrointestinal disorders) | 1 (4)
Pleuritis sicca (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGOS-SC Sensor (N=22)
Cataract (Eye disorders) | 3 (3)
COVID-19 infection (Infections and infestations) | 4 (5)
Increased intraocular pressure (Investigations) | 4 (5)
Increased intraocular pressure -non-study eye- (Investigations) | 2 (2)
Visual acuity reduced (Eye disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT04773106/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT04773106/SAP_001.pdf